CLINICAL TRIAL: NCT06343142
Title: Effects of Time of Day and Nut Intake on Cognitive Performance: a Crossover Trial in Healthy Adults
Brief Title: Effects of Time of Day and Nut Intake on Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Barbara R. Cardoso, Senior Lecturer, Monash University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Nuts for thought
Record Dates: First submitted 2024-03-27; First posted 2024-04-02 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Cognitive Performance
MeSH Terms: interventions — Nuts

STUDY DESIGN:
Intervention Model Description: 2 x 2-factor crossover design study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Lunch nut-free meal (Placebo Comparator): Participants will receive an isocaloric meal without nuts at lunchtime.
  Interventions: Other: Nut-free meal
- Lunch nut meal (Experimental): Participants will receive an isocaloric meal with nuts at lunchtime.
  Interventions: Other: Nuts
- Dinner nut-free meal (Placebo Comparator): Participants will receive an isocaloric meal without nuts at dinner.
  Interventions: Other: Nut-free meal
- Dinner nut meal (Experimental): Participants will receive an isocaloric meal with nuts at dinner.
  Interventions: Other: Nuts

INTERVENTIONS:
Other: Nuts — Isocaloric meal with nuts
  Arms: Dinner nut meal; Lunch nut meal
Other: Nut-free meal — Isocaloric meal without nuts
  Arms: Dinner nut-free meal; Lunch nut-free meal

SUMMARY:
This is a 2 x 2-factor crossover design study to investigate the effects of time of day and nuts on post-meal cognitive performance.

DETAILED DESCRIPTION:
In this trial, eligible participants will receive isocaloric meals with or without nuts at lunchtime and dinner time. Cognitive performance will be performed before and 90 min after the meals.

ELIGIBILITY:
Inclusion Criteria:

* Non-shift workers
* 18-55 years
* BMI between 18.5 and 27 kg/m2,
* Non-smokers
* Without chronic illnesses

Exclusion Criteria:

* Allergy to nuts
* BMI<18.5 or >27 kg/m2
* Presence of dementia or psychiatric disease (depression, Parkinson's disease, schizophrenia)
* Presence of diabetes, serious health conditions that may affect participation e.g. liver or thyroid dysfunction, recent major surgery, cardiovascular disease
* Presence of any sleep disorders
* Taking anti-diabetic or lipid-lowering medication
* Do not speak English
* Pregnant or planning on becoming pregnant
* Breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
N-back task - accuracy | before meal x 90 min post-meal
  Difference in the total accuracy
N-back task - matched responses | before meal x 90 min post-meal
  Difference in the % matched responses
N-back task - false alarm | before meal x 90 min post-meal
  Difference in the % false alarm
N-back task - reaction time | before meal x 90 min post-meal
  Difference in the reaction time for correct matched responses
Stroop test - congruent | before meal x 90 min post-meal
  Difference in the reaction time for congruent
Stroop test - incongruent | before meal x 90 min post-meal
  Difference in the reaction time for incongruent
Stroop test - interference | before meal x 90 min post-meal
  Difference in stroop interference (incongruent - congruent response time)

SECONDARY OUTCOMES:
Multitasking - pure blocks | before meal x 90 min post-meal
  Difference in the reaction time for pure blocks
Multitasking - mixed blocks | before meal x 90 min post-meal
  Difference in the reaction time for mixed blocks
Multitasking - mixing cost | before meal x 90 min post-meal
  Difference in mixing cost (mixed - pure reaction time)
Satiety - hunger | Hunger will be assessed with a visual analog scale before the meal and 4 times after the meal (15, 30, 60 and 90 mins).
  Difference in postprandial hunger
Satiety - fullness | Fullness will be assessed with a visual analog scale before the meal and 4 times after the meal (15, 30, 60 and 90 mins).
  Difference in postprandial fullness
Satiety - satisfaction | Satisfaction will be assessed with a visual analog scale before the meal and 4 times after the meal (15, 30, 60 and 90 mins).
  Difference in postprandial satisfaction
Satiety - eating capacity | Eating capacity will be assessed with a visual analog scale before the meal and 4 times after the meal (15, 30, 60 and 90 mins).
  Difference in postprandial eating capacity,
Satiety index | Satiety index will be assessed before the meal and 4 times after the meal (15, 30, 60 and 90 mins).
  Difference in postprandial satiety index, calculated using the mean of the four satiety questions, where "hunger" and "eating capacity" will be scored in an inverse way than "fullness" and "satisfaction".

CONTACTS AND LOCATIONS:
Overall Officials: Barbara R Cardoso, PhD, Principal Investigator — Department of Nutrition, Dietetics and Food - Monash University; Maxine Bonham, PhD, Principal Investigator — Department of Nutrition, Dietetics and Food - Monash University; Helen Macpherson, PhD, Principal Investigator — Deakin University
Locations (1):
- Department of Nutrition, Dietetics and Food - Monash University, Notting Hill, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No